CLINICAL TRIAL: NCT01397929
Title: An Open-Label Phase I/IIa Study of Intravenous BAL101553 in Adult Patients With Advanced Solid Tumors
Brief Title: An Open-Label Study of Intravenous BAL101553 in Adult Patients With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDI-CS-001
Record Dates: First submitted 2011-07-12; First posted 2011-07-20 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Solid Organ Tumors
MeSH Terms: interventions — lisavanbulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: BAL101553 at MTD (Experimental)
  Interventions: Drug: BAL101553
- Drug: BAL101553 at 50% of MTD (Experimental)
  Interventions: Drug: BAL101553

INTERVENTIONS:
Drug: BAL101553 — Intravenous administration

SUMMARY:
First in human, open-label, sequential dose escalation and expansion study of intravenous BAL101553 in adult patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with one of the following advanced or recurrent solid tumor types, who failed standard therapy or for whom no effective standard therapy is available:colorectal; gastric or cancers of the gastro-esophageal junction; non-small cell lung cancer; ovarian (or primary peritoneal); pancreatic (including ampullary); triple-negative breast
3. Measurable tumor disease (or non-measurable ovarian cancer that can be followed by CA-125)
4. Life expectancy ≥ 12 weeks
5. Acceptable organ and marrow function at baseline (protocol defined laboratory parameters)
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
7. Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

1. Patients who have received chemotherapy, radiotherapy, immunotherapy, or investigational agents within 4 weeks prior to starting study drug or who have not recovered from side effects of prior therapies
2. Symptomatic brain metastases (including leptomeningeal disease) indicative of active disease
3. Peripheral neuropathy ≥ CTCAE v4 grade 2
4. Uncontrolled intercurrent illness that would unduly increase the risk of toxicity or limit compliance with study requirements
5. Women who are pregnant or breast-feeding. Men or women of reproductive potential who are not willing to apply effective birth control
6. Systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg observed as part of the screening examination.
7. Patients treated with a calcium channel blocker or who require combination of more than 2 antihypertensives to control blood pressure.
8. Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-06; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose and characterize dose limiting toxicities of BAL101553 | 28 day cycles
  First-cycle dose limiting toxicities (DLT)

SECONDARY OUTCOMES:
To evaluate safety and tolerability of BAL101553 treatment | 28 day cycles
  Incidence of adverse events, laboratory abnormalities, clinically significant changes in vital signs or ECG assessments
To evaluate BAL101553 pharmacokinetics | 28 day cycles
  BAL101553 and BAL27862 PK parameters including (but not limited to): Cmax (maximum observed plasma concentration), AUC (area under the concentration time curve), half-life, volume of distribution
To assess anti-tumor activity of BAL101553 | 28 day cycles
  Response rate per RECIST guidelines
To explore the use of biomarkers and to characterize pharmacodynamic effects of BAL101553 | 28 day cycles
  Exploratory assessment of baseline levels and change from baseline in the number of circulating tumor cells and other biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, MD, Study Director — Basilea Pharmaceutica International Ltd
Locations (3):
- United Kingdom (3):
  - Royal Marsden Hospital, Sutton, Surrey
  - University College London NHS Foundation Trust, London
  - Sir Bobby Robson Cancer Trials Research Centre; Northern Centre for Cancer Care, Newcastle upon Tyne